CLINICAL TRIAL: NCT03165084
Title: iSMS: Person-centred Interactive Self-management Support in Primary Healthcare for People With Type 2 Diabetes - A Randomized Controlled Trial
Brief Title: Person-centred Interactive Self-management Support in Primary Healthcare for People With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: The Swedish Diabetes Foundation (Unknown); The County Council of Västerbotten (Unknown)
Responsible Party: Principal Investigator, Ulrika Öberg, MSc, PhD student, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iSMS-1
Record Dates: First submitted 2017-05-05; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Type 2
Keywords: Self-management; Primary Health Care; eHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Experimental): Participants in the intervention group will receive usual care, and also use a diabetesapp and a homepage and advice personally tailored according to the personal needs to provide support for them to manage e.g. food choices, exercise, medicine, blood sugars and emotional adaptation.
  Interventions: Behavioral: Intervention arm: Person-centred interactive self-management support
- Control arm (Other): Participants in the control group will receive usual care and also take part in a minimal intervention in the form of a brochure on the importance of self-management in diabetes.
  Interventions: Other: Control arm
- External comparison group (Other): An external comparison group will be recruited from two other primary health care centers in order to analyse possible Hawthorne effects.
  Interventions: Other: External comparison group

INTERVENTIONS:
Behavioral: Intervention arm: Person-centred interactive self-management support — Person-centred tailored digital self-management support hypothesised to decrease HbA1c, improve other metabolic measurements, improve lifestyle habits, and increase diabetes empowerment, increase diabetes-dependent quality of life, improve illness perception, and improve eHealth literacy.
  Access to the diabetes mobile application and the homepage during 16 weeks. Each individual will set personal goals for use of the digital resources.
  Arms: Intervention arm
Other: Control arm — Participants will receive usual care and take part in a minimal intervention in the form of a brochure on the importance of self-management in diabetes.
  Arms: Control arm
Other: External comparison group — External comparison groups in order to analyse possible Hawthorne effects.
  Arms: External comparison group

SUMMARY:
The aim of this study is to develop and evaluate a person-centred digital intervention in primary healthcare for people with T2D, in addition to their usual diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes within the last five years
* 18 years of age or older
* Ability to read and communicate in Swedish
* Own a smart phone

Exclusion Criteria:

* 81 years and over at inclusion
* Life-threatening physical illness (e.g. cancer)
* Documented cognitive impairment
* Those not responsible for their own self care
* Those not residing in their own home environment (e.g. those in nursing homes, in-patient hospital wards)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, 6 months, and 12 months
  Change from baseline in HbA1c at 6 months and 1 year (in mmol/mol)

SECONDARY OUTCOMES:
Systolic blood pressure | Baseline, 6 months, and 12 months
  Change from baseline in systolic blood pressure at 6 months and 1 year
Body Mass Index | Baseline, 6 months, and 12 months
  Change from baseline in Body Mass Index at 6 months and 1 year
Waist circumference | Baseline, 6 months, and 12 months
  Change from baseline in waist circumference at 6 months and 1 year
Cholesterol, total, LDL and HDL | Baseline, 6 months, and 12 months
  Change from baseline in Cholesterol, total, LDL and HDL at 6 months and 1 year
Lifestyle habits - physical activity | Baseline, 6 months, and 12 months
  Change from baseline in lifestyle habits - physical activity via questionnaires at 6 months and 1 year
Lifestyle habits - diet | Baseline, 6 months, and 12 months
  Change from baseline in lifestyle habits - diet via questionnaires at 6 months and 1 year
Lifestyle habits - smoking | Baseline, 6 months, and 12 months
  Change from baseline in lifestyle habits - smoking via questionnaires at 6 months and 1 year
Medical treatment | Baseline, 6 months, and 12 months
  Change in the drug dosage from baseline in medical treatment via questionnaires at 6 months and 1 year
Diabetes empowerment | Baseline, 6 months, and 12 months
  Change from baseline in diabetes empowerment via questionnaires at 6 months and 1 year
Diabetes-dependent QoL | Baseline, 6 months, and 12 months
  Change from baseline in diabetes-dependent QoL at 6 months and 1 year
Illness perception | Baseline, 6 months, and 12 months
  Change from baseline in illness perception via questionnaires at 6 months and 1 year
eHealth literacy | Baseline, 6 months, and 12 months
  Change from baseline in eHealth literacy at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Hörnsten, Professor, Study Director — Umeå University
Locations (1):
- Department of Nursing, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No